CLINICAL TRIAL: NCT02629822
Title: A Phase IIa Multicenter, Open-Label Clinical Trial to Evaluate the Safety and Efficacy of MK-1439A in Treatment-Naïve HIV-1 Infected Subjects With Selected Non-Nucleoside Reverse Transcriptase Inhibitor (NNRTI) Transmitted Resistance Mutations
Brief Title: Safety and Efficacy of Doravirine, Tenofovir, Lamivudine (MK-1439A) in Participants Infected With Treatment-Naïve Human Immunodeficiency Virus (HIV) -1 With Transmitted Resistance (MK-1439A-030)
Acronym: DRIVE BEYOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1439A-030; 2015-003616-20 (EudraCT Number); MK-1439A-030 (Other: Merck)
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DOR/3TC/TDF (Experimental): Treatment-naïve HIV-1 infected participants with NNRTI transmitted resistance-associated mutations were treated with open-label MK-1439A (DOR/3TC/TDF 100mg/300mg/300mg) as a FDC tablet taken once daily by mouth for 96 weeks in the Base Study. In addition, eligible participants continued to receive the same MK-1439A regimen from Week 96 to Week 192 during the Extension Study.
  Interventions: Drug: Doravirine/lamivudine/tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Doravirine/lamivudine/tenofovir disoproxil fumarate — FDC tablet containing MK-1439 (doravirine) 100 mg / lamivudine 300 mg / tenofovir disoproxil fumarate 300 mg taken by mouth.
  Other Names: MK-1439A; DELSTRIGO™

SUMMARY:
The primary objectives of this study are to evaluate the antiretroviral activity and the safety/tolerability of open-label doravirine/lamivudine/tenofovir disoproxil fumarate (DOR/3TC/TDF; MK-1439A; DELSTRIGO™) consisting of a single fixed-dose combination (FDC) tablet of DOR/3TC/TDF 100 mg/300 mg/300 mg in treatment-naïve HIV-1 infected participants with select non-nucleoside reverse transcriptase inhibitor (NNRTI) transmitted resistance-associated mutations.

DETAILED DESCRIPTION:
This study had a Base Study (Day 1 to Week 96) and an optional Study Extension (Week 96 to Week 192).

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive within 45 days prior to the treatment phase of this study, and have HIV treatment indicated based on physician assessment.
* Is naïve to antiretroviral therapy (ART) including investigational antiretroviral agents.
* Prior to screening, have had a genotype performed confirming the presence of only one of the following NNRTI mutations: K103N, Y181C, or G190A.
* Is considered clinically stable with no signs or symptoms of active infection at time of entry into the study (i.e. clinical status and all chronic medications should be unchanged for at least 2 weeks prior to the start of treatment in this study).
* Is highly unlikely to become pregnant or to impregnate a partner

Exclusion Criteria:

* Is a user of recreational or illicit drugs or has had a recent history of drug or alcohol abuse or dependence.
* Has been treated for a viral infection other than HIV-1, such as hepatitis B, with an agent that is active against HIV-1, including, but not limited to, adefovir, tenofovir, entecavir, emtricitabine, or lamivudine.
* Has documented or known resistance to study drugs (doravirine, lamivudine, and/or tenofovir)
* Has participated or anticipates participating in a study with an investigational compound/device within 30 days prior to signing informed consent
* Has any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppressant drugs during the course of the trial.
* Requires or anticipates requiring any of the prohibited medications
* Has significant hypersensitivity or other contraindication to any of the components of the study drug
* Has a current (active) diagnosis of acute hepatitis due to any cause
* Has evidence of decompensated liver disease or has liver cirrhosis and a Child-Pugh Class C score or Pugh-Turcotte (CPT) score > 9
* Is pregnant, breastfeeding, or expecting to conceive
* Is female and expecting to donate eggs, or is male and is expecting to donate sperm at any time during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wong A, Goldstein D, Mallolas J, DeJesus E, Johnson M, Molina JM, Pozniak A, Rodgers A, Teal V, Hepler D, Kumar S, Sklar P, Hanna GJ, Hwang C, Badshah C, Teppler H. Efficacy and Safety of Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate (DOR/3TC/TDF) in Treatment-Naive Adults With HIV-1 and Transmitted Nonnucleoside Reverse Transcriptase Inhibitor Resistance Mutations. J Acquir Immune Defic Syndr. 2019 Dec 1;82(4):e47-e49. doi: 10.1097/QAI.0000000000002153. PMID 31425317

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 7 study sites in Canada, France, Spain, UK, and USA.
Groups:
- DOR/3TC/TDF: Treatment-naïve HIV-1 infected participants with NNRTI transmitted resistance-associated mutations were treated with open-label MK-1439A (DOR/3TC/TDF 100mg/300mg/300mg) as a FDC tablet taken once daily by mouth for 96 weeks in the Base Study. In addition, eligible participants continued to receive the same MK-1439A regimen from Week 96 to Week 192 during the optional Extension Study.
Period: Base Study
Arm/Group | DOR/3TC/TDF
Started | 10
Completed | 7
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Non-Compliance With Study Drug | 1
Period: Extension Study
Arm/Group | DOR/3TC/TDF
Started | 6 (Enrollment in Extension Study was voluntary.)
Completed | 4
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (32.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving HIV-1 Ribonucleic Acid (RNA) <50 Copies/mL of Plasma at Week 48
Description: The percentage of participants achieving HIV-1 ribonucleic acid (RNA) <50 copies/mL in plasma at Week 48 was calculated. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification (LoQ) of 40 copies/mL, was used to measure the HIV-1 RNA level in plasma samples obtained at Week 48 visit.
Time Frame: Week 48
Population: All participants who received ≥1 dose of MK-1439A, had baseline and Week 48 data for HIV in plasma, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 8
Percentage of Participants | 100.0 [63.1 to 100.0]

2. Primary Outcome: Percentage of Participants Experiencing ≥1 Adverse Events (AE) up to Week 48
Description: The percentage of participants experiencing ≥1 AE up to Week 48 was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to Week 48
Population: All participants who received ≥1 dose of MK-1439A.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 10
Percentage of Participants | 90.0

3. Primary Outcome: Percentage of Participants Who Discontinued Treatment Due to an AE up to Week 48.
Description: The percentage of participants who discontinued from study medication due to an adverse event was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to Week 48
Population: All participants who received ≥1 dose of MK-1439A.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 10
Percentage of Participants | 0.0

4. Primary Outcome: Percentage of Participants Experiencing ≥1 Adverse Events (AE) up to Week 96
Description: The percentage of participants experiencing ≥1 AE up to Week 96 was calculated. An AE was defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy could be determined.
Time Frame: Up to Week 96
Population: All participants who received ≥1 dose of MK-1439A.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 10
Percentage of Participants | 90.0

5. Primary Outcome: Percentage of Participants Who Discontinued Treatment Due to an AE up to Week 96
Description: as for outcome 3
Time Frame: Up to Week 96
Population: All participants who received ≥1 dose of MK-1439A.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 10
Percentage of Participants | 0.0

6. Secondary Outcome: Percentage of Participants Achieving HIV-1 Ribonucleic Acid (RNA) <50 Copies/mL of Plasma at Week 96
Description: The percentage of participants achieving HIV-1 ribonucleic acid (RNA) <50 copies/mL in plasma at Week 96 was calculated. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification (LoQ) of 40 copies/mL, was used to measure the HIV-1 RNA level in plasma samples obtained at Week 96 visit.
Time Frame: Week 96
Population: All participants who received ≥1 dose of MK-1439A, had baseline and Week 96 data for HIV in plasma, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 7
Percentage of Participants | 100.0 [59.0 to 100.0]

7. Secondary Outcome: Percentage of Participants Achieving HIV-1 Ribonucleic Acid (RNA) <40 Copies/mL of Plasma at Week 48
Description: The percentage of participants achieving HIV-1 ribonucleic acid (RNA) <40 copies/mL in plasma at Week 48 was calculated. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification (LoQ) of 40 copies/mL, was used to measure the HIV-1 RNA level in plasma samples obtained at Week 48 visit. Participants with reading below the LoQ were considered to have <40 copies/mL.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 8
Percentage of Participants | 100.0 [63.1 to 100.0]

8. Secondary Outcome: Percentage of Participants Achieving HIV-1 Ribonucleic Acid (RNA) <40 Copies/mL of Plasma at Week 96
Description: The percentage of participants achieving HIV-1 ribonucleic acid (RNA) <40 copies/mL in plasma at Week 96 was calculated. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification (LoQ) of 40 copies/mL, was used to measure the HIV-1 RNA level in plasma samples obtained at Week 96 visit. Participants with reading below the LoQ were considered to have <40 copies/mL.
Time Frame: Week 96
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 7
Percentage of Participants | 100.0 [59.0 to 100.0]

9. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Description: The change from baseline in CD4 cell count at Week 48 was calculated.
Time Frame: Baseline (Day 1) and Week 48
Population: All participants who received ≥1 dose of MK-1439A, had baseline and Week 48 data for CD4 cell count, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations.
Measure: Mean (95% Confidence Interval); unit: Cells/mm^3
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 8
Cells/mm^3
  Baseline for the Week 48 Population | 409 [293.5 to 525.0]
  Change from Baseline at Week 48 | 132 [24.4 to 239.8]

10. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Description: The change from baseline in CD4 cell count at Week 96 was calculated.
Time Frame: Baseline (Day 1) and Week 96
Population: All participants who received ≥1 dose of MK-1439A, had baseline and Week 96 data for CD4 cell count, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations.
Measure: Mean (95% Confidence Interval); unit: Cells/mm^3
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 7
Cells/mm^3
  Baseline for the Week 96 Population | 437 [323.9 to 550.7]
  Change from Baseline at Week 96 | 153 [23.0 to 282.8]

11. Secondary Outcome: Time to Loss of Virologic Response
Description: The time to loss of virologic response (TLOVR) was reported. For participants who achieved HIV-1 RNA <50 copies/mL of plasma and subsequently had two consecutive HIV-1 RNA values of ≥50 copies/mL measured at least 1 week apart, TLOVR was the time between Day 1 and the date of the first of the two consecutive values ≥50 copies/mL. For participants who achieved and sustained HIV-1 RNA <50 copies/mL, time to loss of virologic response was censored at the time of the last available measurement.
Time Frame: Up to Week 96
Population: All participants who experienced protocol-defined virologic failure, received ≥1 dose of MK-1439A, had baseline and later data for HIV in plasma, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations. Participants who did not experience virologic failure were excluded from the analysis population.
Measure: Mean (Full Range); unit: Days
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 1
Days | 166 [166 to 166]

12. Other Pre Specified Outcome: Percentage of Participants Achieving HIV-1 Ribonucleic Acid (RNA) <50 Copies/mL of Plasma at Week 192
Description: The percentage of participants achieving HIV-1 ribonucleic acid (RNA) <50 copies/mL in plasma at Week 192 was calculated. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification (LoQ) of 40 copies/mL, was used to measure the HIV-1 RNA level in plasma samples obtained at Week 192 visit.
Time Frame: Week 192
Population: All participants who received ≥1 dose of MK-1439A, had baseline and Week 192 data for HIV in plasma, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 4
Percentage of Participants | 100.0 [39.8 to 100.0]

13. Other Pre Specified Outcome: Percentage of Participants Achieving HIV-1 Ribonucleic Acid (RNA) <40 Copies/mL of Plasma at Week 192
Description: The percentage of participants achieving HIV-1 ribonucleic acid (RNA) <40 copies/mL in plasma at Week 192 was calculated. The Abbott RealTime HIV-1 Assay, which has a lower limit of reliable quantification (LoQ) of 40 copies/mL, was used to measure the HIV-1 RNA level in plasma samples obtained at Week 192 visit. Participants with reading below the LoQ were considered to have <40 copies/mL.
Time Frame: Week 192
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 4
Percentage of Participants | 100.0 [39.8 to 100.0]

14. Other Pre Specified Outcome: Change From Baseline in CD4 Cell Count at Week 192
Description: The change from baseline in CD4 cell count at Week 192 was calculated.
Time Frame: Baseline (Day 1) and Week 192
Population: All participants who received ≥1 dose of MK-1439A, had baseline and Week 192 data for CD4 cell count, and whose central lab results confirmed the presence of protocol-specified NNRTI transmitted resistance-associated mutations.
Measure: Mean (95% Confidence Interval); unit: Cells/mm^3
Arm/Group | DOR/3TC/TDF
Number analyzed (Participants) | 4
Cells/mm^3
  Baseline for the Week 192 Population | 479 [310.0 to 648.5]
  Change from Baseline at Week 192 | 196 [27.4 to 364.1]

ADVERSE EVENTS:
Time Frame: Up to 192 Weeks
Description: All participants who received ≥1 dose of study intervention are included in AE results. All-cause mortality is based on all randomized participants.
Groups:
- DOR/3TC/TDF Base Study: Day 1 to Week 96: Treatment-naïve HIV-1 infected participants with NNRTI transmitted resistance-associated mutations were treated with open-label MK-1439A (DOR/3TC/TDF 100mg/300mg/300mg) as a FDC tablet taken once daily by mouth for 96 weeks in the Base Study.
- DOR/3TC/TDF Study Extension: Week 97 to Week 192: Eligible participants who chose to continue on study received the same MK-1439A regimen from Week 96 to Week 192 during the Extension Study.
Arm/Group | DOR/3TC/TDF Base Study: Day 1 to Week 96 | DOR/3TC/TDF Study Extension: Week 97 to Week 192
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 9/10 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/3TC/TDF Base Study: Day 1 to Week 96 (N=10) | DOR/3TC/TDF Study Extension: Week 97 to Week 192 (N=6)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/3TC/TDF Base Study: Day 1 to Week 96 (N=10) | DOR/3TC/TDF Study Extension: Week 97 to Week 192 (N=6)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anogenital dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal tract irritation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gonorrhoea (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis syphilitic (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (5) | 1 (2)
Oropharyngeal gonococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 1 (1) | 0 (0)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Penile discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication (or after public disclosure of the results at www.clinicaltrials.gov if multicenter manuscript is not planned), an investigator and colleagues may publish their data independently. Sponsor must have opportunity to review proposed abstracts, manuscripts or presentations 45 days prior to submission for publication/presentation. Confidential information must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT02629822/Prot_SAP_000.pdf